CLINICAL TRIAL: NCT00755469
Title: Modification of Reperfusion by "Post-Conditioning" Reduces Infarct Size in Acute Myocardial Infarction
Brief Title: Post-conditioning to Reduce Infarct Size
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Society for Cardiovascular Angiography and Interventions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: opt002
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Myocardial Infarction
Keywords: Reperfusion injury; Post-Conditioning; Infarct size
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Post-conditioning

INTERVENTIONS:
Procedure: Post-conditioning — The post-conditioning protocol consists of performing 4, 30-second PTCA balloon occlusions followed by 30 seconds of reperfusion for a total of 4 minutes. The first balloon inflation occurs immediately after an angioplasty guidewire is placed through the obstruction in the artery and flow is restored. Following this protocol the vessel will be stented as part of usual practice for treatment of acute MI.

SUMMARY:
When angioplasty (PTCA) and stenting of the blood vessels of the heart is the treatment for a Heart Attack, there is damage to the heart muscle that is caused by the sudden opening of the blood vessels. This is called "reperfusion injury". The cell death is due to inflammation and the generation of free radicals.

The primary objective of this study is to determine if post-conditioning(four brief (30 second) PTCA balloon inflations) reduces damage to the heart muscle. This will be measured by heart enzyme tests-CK measurements- and by cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 < 80
* Able to give informed consent
* 100% occlusion of a major epicardial vessel with TIMI 0 Flow

Exclusion Criteria:

* Significant collateral blood flow to the distal vasculature of the occluded vessel.
* Previous CABG
* Previous q-wave myocardial infarction in the same territory

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Infarct size, determined by late-enhancement measurements of the LV using gadolinium contrast with cardiac MRI | 3 months

SECONDARY OUTCOMES:
The degree of Microvascular Obstruction (MVO), as measured by Cardiac MRI | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay H Traverse, MD, Principal Investigator — Minneapolis Heart Institute at Abbott Northwestern Hospital
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Traverse JH, Wang YL, Chavez, IJ, Lesser JR, Pedersen WR, Mirheydar H, Henry TD. Post Conditioning reduces infarct size and improves LV function during acute myocardial infarction. Circulation 2006;114:II-344.
- [Background] Staat P, Rioufol G, Piot C, Cottin Y, Cung TT, L'Huillier I, Aupetit JF, Bonnefoy E, Finet G, Andre-Fouet X, Ovize M. Postconditioning the human heart. Circulation. 2005 Oct 4;112(14):2143-8. doi: 10.1161/CIRCULATIONAHA.105.558122. Epub 2005 Sep 26. PMID 16186417
- [Result] Garcia S, Henry TD, Wang YL, Chavez IJ, Pedersen WR, Lesser JR, Shroff GR, Moore L, Traverse JH. Long-term follow-up of patients undergoing postconditioning during ST-elevation myocardial infarction. J Cardiovasc Transl Res. 2011 Feb;4(1):92-8. doi: 10.1007/s12265-010-9252-0. Epub 2010 Dec 7. PMID 21136310
- See also: The Minneapolis Heart Institute Foundation improves cardiovascular health through clinical research and education — http://www.mplsheart.org